CLINICAL TRIAL: NCT04092530
Title: Linking Inter-professional Newborn and Contraception Care (LINCC) Trial - A Novel Approach to Postpartum Contraception Provision at the Well-Baby Visit
Brief Title: Linking Inter-professional Newborn and Contraception Care
Acronym: LINCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Illinois at Chicago (Other); AllianceChicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R01HD097171 (NIH)
Record Dates: First submitted 2019-09-09; First posted 2019-09-17 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Family Planning; Contraception; PostPartum

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation Hybrid Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Aim 2 (Experimental): During the intervention period, staff will capture women during the first well-baby visit (WBV) and offer to have the next visit co-scheduled for infant and contraception care. Appointments are scheduled during the discharge process at the end of each WBV. During the discharge process all women 0-6 months postpartum will be identified by clerical staff through review of each pediatric clinic beforehand and through an electronic flag alert in the infant's electronic medical record. The pre-review of pediatric clinic schedules and the use of the flag will remind staff to offer the mother a co-scheduled visit for newborn and contraceptive care at the time of the next newborn visit.
  Interventions: Behavioral: LINCC intervention - enable co-schedule feature
- Control - Aim 2 (No Intervention): Clinics will schedule postpartum contraception using normal clinic procedures.

INTERVENTIONS:
Behavioral: LINCC intervention - enable co-schedule feature — Clinics will offer postpartum contraception appointments earlier and the opportunity to co-schedule these appointments with their infant's next well-baby visit
  Arms: Intervention - Aim 2

SUMMARY:
Pregnancies conceived within 18 months of a prior delivery (termed short inter-pregnancy interval [IPI]) place mothers and infants at high risk for poor health outcomes and affect nearly one third of women in the U.S. Rates of postpartum (PP) contraception use remain low, particularly among low-income minority women, leading to high rates of short IPI pregnancies. This proposed study aims to address the gap in the current model of PP contraception care, by developing and implementing a novel approach to link (co-schedule) PP contraception care with newborn well-baby care with the goal of improving access to timely PP contraception.

DETAILED DESCRIPTION:
Pregnancies conceived within 18 months of a prior delivery (termed short inter-pregnancy interval [IPI]) place mothers and infants at high risk for poor health outcomes including pre-eclampsia, anemia, and preterm birth. Despite these negative health consequences, nearly one third of women experience a short IPI, highlighting a significant public health problem in the U.S. A critical approach to preventing short IPIs is to provide postpartum (PP) women with timely access to contraception. The current standard clinical practice is to have women return six weeks after delivery for a postpartum visit, at which time contraceptive needs are addressed. However, many women resume sexual activity prior to six weeks PP, and many women, particularly low-income minority women, do not present for this visit. Low rates of postpartum contraception uptake leave women vulnerable to an unplanned pregnancy and significant negative health consequences. Thus, there is an urgent need for alternative approaches to increase timely access to PP contraception to improve outcomes for women and children.

The proposed study aims to:

1. develop a comprehensive implementation plan to link PP contraception and newborn care through co-scheduling visits in community health centers (CHC);
2. use an effectiveness- implementation hybrid design to evaluate this novel system-level approach to linking maternal and newborn care at CHCs served by our partner organization, AllianceChicago and;
3. assess implementation of linked PP contraception and newborn care and report on key barriers and facilitators related to successful implementation of the intervention.

Increasing access to timely contraception is a promising strategy to help women plan their families and, in turn, reduce the poor health sequela associated with short IPI pregnancies. The long-term impact of this study is to reduce negative health outcomes among PP women and infants by increasing access to patient-oriented PP contraceptive care. Findings may provide evidence supporting a paradigm shift for linked PP care and identify important insights to facilitate successful implementation of this model of care in CHCs across the nation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants include women presenting with their infants at one of the 7 chosen CHC sites for their first WBV (typically 3-5 days after delivery).

Exclusion Criteria:

* Women will be excluded if they had a tubal ligation or a long acting reversible contraception planned immediately after delivery. Additionally, women will be excluded if they needed an emergency hysterectomy due to life threatening bleeding during delivery. Any male patients will be excluded from the study because the study outcomes of contraceptive method use and pregnancy status are not applicable to males.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2518 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Haider, MD, Principal Investigator — Rush University Medical Center; Rachel Caskey, MD, Principal Investigator — University of Illinois at Chicago
Locations (5):
- United States (5):
  - Malama O ke Ola, Wailuku, Hawaii
  - Friend Health, Chicago, Illinois
  - Heartland Health Centers, Chicago, Illinois
  - Infant Welfare Society, Chicago, Illinois
  - Settlement Health, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed at the Community Health Clinic (CHC) level in this cluster-randomized trial, so all eligible patients at each CHC were included in the analysis of outcome data. No individual patient recruitment was performed.
Pre-assignment Details: Seven CHCs were enrolled and all eligible patients from those CHCs were included in the outcome assessment. Randomization occurred at the CHC level, then the stepped wedge design was applied to roll out the intervention in waves according to the sequence. Therefore, patients seen at any given CHC prior to the implementation of the intervention were assigned to the Control condition and those seen at that CHC after the implementation of the intervention were assigned to the Intervention condition
Units Other Than Participants: Clinics
Groups:
- Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention: Clinic 1 was randomly assigned to start the clinic-level intervention after 3 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 21 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention: Clinic 2 was randomly assigned to start the clinic-level intervention after 6 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 18 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention: Clinic 3 was randomly assigned to start the clinic-level intervention after 9 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 15 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention: Clinic 4 was randomly assigned to start the clinic-level intervention after 12 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 12 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention: Clinic 5 was randomly assigned to start the clinic-level intervention after 15 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 9 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention: Clinic 6 was randomly assigned to start the clinic-level intervention after 18 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 6 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
- Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention: Clinic 7 was randomly assigned to start the clinic-level intervention after 21 months in the baseline period followed by 3 months for training and wash out. The intervention period continued for 3 months at this clinic. During the intervention period, staff approached women during all well-baby visits (WBV) between 0-6 months and offered to have the next visit co-scheduled for infant and contraception care. Appointments were scheduled during the discharge process at the end of each WBV.
Period: Period 1: Months 1-3
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 82; 1 Clinics | 50; 1 Clinics | 68; 1 Clinics | 32; 1 Clinics | 52; 1 Clinics | 17; 1 Clinics | 12; 1 Clinics
Completed | 82; 1 Clinics | 50; 1 Clinics | 68; 1 Clinics | 32; 1 Clinics | 52; 1 Clinics | 17; 1 Clinics | 12; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 2: Months 4-6
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 0; 0 Clinics (Training/Washout period) | 36; 1 Clinics | 74; 1 Clinics | 42; 1 Clinics | 50; 1 Clinics | 31; 1 Clinics | 13; 1 Clinics
Completed | 0; 0 Clinics | 36; 1 Clinics | 74; 1 Clinics | 42; 1 Clinics | 50; 1 Clinics | 31; 1 Clinics | 13; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 3: Months 7-9
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 78; 1 Clinics | 0; 0 Clinics (Training/Washout period) | 74; 1 Clinics | 29; 1 Clinics | 59; 1 Clinics | 30; 1 Clinics | 15; 1 Clinics
Completed | 78; 1 Clinics | 0; 0 Clinics | 74; 1 Clinics | 29; 1 Clinics | 59; 1 Clinics | 30; 1 Clinics | 15; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 4: Months 10-12
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 65; 1 Clinics | 42; 1 Clinics | 0; 0 Clinics (Training/Washout period) | 48; 1 Clinics | 46; 1 Clinics | 24; 1 Clinics | 19; 1 Clinics
Completed | 65; 1 Clinics | 42; 1 Clinics | 0; 0 Clinics | 48; 1 Clinics | 46; 1 Clinics | 24; 1 Clinics | 19; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 5: Months 13-15
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 60; 1 Clinics | 48; 1 Clinics | 83; 1 Clinics | 0; 0 Clinics (Training/Washout period) | 39; 1 Clinics | 25; 1 Clinics | 11; 1 Clinics
Completed | 60; 1 Clinics | 48; 1 Clinics | 83; 1 Clinics | 0; 0 Clinics | 39; 1 Clinics | 25; 1 Clinics | 11; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 6: Months 16-18
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 46; 1 Clinics | 48; 1 Clinics | 91; 1 Clinics | 47; 1 Clinics | 0; 0 Clinics | 27; 1 Clinics | 6; 1 Clinics
Completed | 46; 1 Clinics | 48; 1 Clinics | 91; 1 Clinics | 47; 1 Clinics | 0; 0 Clinics | 27; 1 Clinics | 6; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 7: Months 19-21
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 66; 1 Clinics | 55; 1 Clinics | 82; 1 Clinics | 29; 1 Clinics | 39; 1 Clinics | 0; 0 Clinics (Training/Washout period) | 10; 1 Clinics
Completed | 66; 1 Clinics | 55; 1 Clinics | 82; 1 Clinics | 29; 1 Clinics | 39; 1 Clinics | 0; 0 Clinics | 10; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 8: Months 22-24
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 76; 1 Clinics | 69; 1 Clinics | 74; 1 Clinics | 29; 1 Clinics | 28; 1 Clinics | 24; 1 Clinics | 0; 0 Clinics (Training/Washout period)
Completed | 76; 1 Clinics | 69; 1 Clinics | 74; 1 Clinics | 29; 1 Clinics | 28; 1 Clinics | 24; 1 Clinics | 0; 0 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics
Period: Period 9: Months 25-27
Arm/Group | Sequence/Clinic 1: 3 Months Baseline, 21 Months Intervention | Sequence/Clinic 2: 6 Months Baseline, 18 Months Intervention | Sequence/Clinic 3: 9 Months Baseline, 15 Months Intervention | Sequence/Clinic 4: 12 Months Baseline, 12 Months Intervention | Sequence/Clinic 5: 15 Months Baseline, 9 Months Intervention | Sequence/Clinic 6: 18 Months Baseline, 6 Months Intervention | Sequence/Clinic 7: 21 Months Baseline, 3 Months Intervention
Started | 71; 1 Clinics | 57; 1 Clinics | 75; 1 Clinics | 38; 1 Clinics | 48; 1 Clinics | 19; 1 Clinics | 10; 1 Clinics
Completed | 71; 1 Clinics | 57; 1 Clinics | 75; 1 Clinics | 38; 1 Clinics | 48; 1 Clinics | 19; 1 Clinics | 10; 1 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Seven control participants had invalid values for age after calculating from their dates of birth, so were not analyzed for the age measure only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Aim 2 | Control - Aim 2 | Total
Number analyzed (Participants) | 1497 | 1021 | 2518
Age, Categorical [Count of Participants; unit: Participants] — Population: Seven control participants had invalid values for age after calculating from their dates of birth, so were not analyzed for the age measure .
  Participants
    number analyzed (Participants) | 1497 | 1014 | 2511
    <=18 years | 44 | 42 | 86
    Between 18 and 65 years | 1453 | 972 | 2425
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Seven control participants had invalid values for age after calculating from their dates of birth, so were not analyzed for the age measure . Population: Seven control participants had invalid values for age after calculating from their dates of birth, so were not analyzed for the age measure .
  years
    number analyzed (Participants) | 1497 | 1014 | 2511
    (all) | 28.5 (6.0) | 27.8 (6.0) | 28.2 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1497 | 1021 | 2518
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1497 | 1021 | 2518
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 70 | 29 | 99
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 551 | 266 | 817
  White | 569 | 547 | 1116
  More than one race | 202 | 129 | 331
  Unknown or Not Reported | 105 | 50 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 438 | 490 | 928
  Not Hispanic or Latino | 954 | 481 | 1435
  Unknown or Not Reported | 105 | 50 | 155

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Receive Contraception by Two Months Postpartum
Description: Using de-identified patient data collected through clinic's Electronic Health Record (EHR) system (i.e., visit type attended, billing codes for contraception) we will measure receipt of all methods of contraception by two months postpartum
Time Frame: 2 months
Population: No difference
Measure: Number; unit: Participants
Units Other Than Participants: Community Health Clinics (CHC)
Arm/Group | Intervention - Aim 2 | Control - Aim 2
Number analyzed (Participants) | 1497 | 1021
Number analyzed (Community Health Clinics (CHC)) | 7 | 7
Participants | 474 | 339
Statistical Analysis 1: Comparison: Intervention - Aim 2 vs Control - Aim 2; Please note that there were only 7 units (community health clinics) analyzed at Level 2 of this multilevel study, but due to the crossover design of the study, they were each observed under both the Control and Intervention conditions. Therefore, the Units Analyzed entered above reflect the 7 clinics under both conditions and should not be summed to 14; Test type: Other; p = 0.12, Mixed Models Analysis; Adjusted for time; clustering by clinical site accounted for with random intercept; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.64 to 1.05]

2. Secondary Outcome: Number of Patients Who Receive Contraception by Six Months Postpartum
Description: Using de-identified patient data collected through clinic's Electronic Medical Record system (i.e., visit type attended, billing codes for contraception) we will measure receipt of all methods of contraception by six months postpartum
Time Frame: 6 months
Population: The stepped wedge design was interrupted for outcomes measured at six months due to a longer washout period, resulting in slightly different, yet overlapping samples for the primary and secondary outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Aim 2 | Control - Aim 2
Number analyzed (Participants) | 1461 | 1067
Participants | 595 | 436
Statistical Analysis 1: Comparison: Intervention - Aim 2 vs Control - Aim 2; Test type: Other; p = 0.33, Mixed Models Analysis; Adjusted for time; random intercept for clinical site; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.70 to 1.13]

3. Secondary Outcome: Number of Patients Who Present With a Short Inter-pregnancy Interval Pregnancies
Description: Use EHR data to follow up participants for short IPI (subsequent pregnancy before 12 months postpartum)
Time Frame: 12 months
Population: Due to a shortened study period because of interruptions related to the COVID-19 pandemic, this outcome was measured at 12 instead of 18 months postpartum. Two clinical sites changed to a new EHR platform before the end of the 12 month follow up period, disrupting follow up and leading to fewer numbers of participants in the intervention condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Aim 2 | Control - Aim 2
Number analyzed (Participants) | 991 | 1067
Participants | 67 | 55
Statistical Analysis 1: Comparison: Intervention - Aim 2 vs Control - Aim 2; Test type: Other; p = 0.88, Mixed Models Analysis; Adjusted for time; random intercept for clinical site; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.33 to 3.73]

ADVERSE EVENTS:
Time Frame: up to 12 months
Groups:
- Experimental: Intervention - Aim 2: During the intervention period, staff will capture women during the first well-baby visit (WBV) and offer to have the next visit co-scheduled for infant and contraception care. Appointments are scheduled during the discharge process at the end of each WBV. During the discharge process all women 0-6 months postpartum will be identified by clerical staff through review of each pediatric clinic beforehand and through an electronic flag alert in the infant's electronic medical record. The pre-review of pediatric clinic schedules and the use of the flag will remind staff to offer the mother a co-scheduled visit for newborn and contraceptive care at the time of the next newborn visit.
Arm/Group | Experimental: Intervention - Aim 2 | Control - Aim 2
All-Cause Mortality (participants affected / at risk) | 0/1497 | 0/1021
Serious Adverse Events (participants affected / at risk) | 0/1497 | 0/1021
Other Adverse Events (participants affected / at risk) | 0/1497 | 0/1021

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04092530/Prot_SAP_000.pdf